CLINICAL TRIAL: NCT02412748
Title: African American Non-Resident Fatherhood Program: Effects on Child/Family Outcomes
Brief Title: The Dedicated African American Dad Study
Acronym: DAAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Wrenetha Julion, Professor, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2R01NR011182-03 (NIH); 2R01NR011182-03 (NIH)
Record Dates: First submitted 2015-03-06; First posted 2015-04-09 (Estimated); Results first posted 2023-04-20 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Father - Child Relations
Keywords: Non-Resident; Fathers; African American

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Financial Literacy Program (Active Comparator): The Financial Literacy Program (FLP) attention control condition will not receive any information on fatherhood. They will participate in a nine-session financial education program, called "Money Smart," which has modules that will be facilitated by a group leader that focus on banking, borrowing, checking accounts, money management, saving, establishing and repairing a credit history, using credit cards responsibly and learning about borrowing and home ownership. They will also receive a booster session 6 weeks after the final session that focuses on setting financial goals.
  Interventions: Behavioral: Financial Literacy Program
- BBTF Intervention (Experimental): The Building Bridges to Fatherhood (BBTF) intervention employs the following key features: a collaborative model for working with parents; vignettes of father-child models engaged in situations typical of non-resident fathers with young children for stimulating discussion and problem-solving; group discussion format, which allows fathers to support one another and share ideas on using program principles to fit within the contexts of fatherhood; "homework assignments" that help fathers practice the new skills at home; weekly handouts summarizing the major points discussed each week, which can be shared with others and used to gain greater support from extended family; and a Leader's Manual that standardizes the program across groups and group leaders.
  Interventions: Behavioral: BBTF Intervention

INTERVENTIONS:
Behavioral: BBTF Intervention — The Building Bridges to Fatherhood (BBTF) intervention consists of 9 group sessions and 1 booster session as described in the arm/group descriptions.
  Arms: BBTF Intervention
Behavioral: Financial Literacy Program — The Financial Literacy Program (FLP) attention control condition consists of 9 group sessions and 1 booster session as described in the arm/group descriptions.
  Arms: Financial Literacy Program

SUMMARY:
The number of children living apart from their fathers has grown nationally, and the greatest percentage is evident among African American (AA) families; two-thirds of all African American children live in households without their biological father. Research supports the importance of positive fathering in the lives of children. But in order for children to benefit from their fathers' involvement, the father-child relationship must be timely and sustained. This study will test culturally relevant interventions aimed at increasing non-resident (not living with the child) AA fathers' involvement with their children.

DETAILED DESCRIPTION:
The purpose of this competing continuation study is to test the efficacy of the core 9-session BBTF program (held over12-weeks) on: (1) improving father outcomes (psychological well-being, relationship quality with the child's mother, parenting competence); (2) father-mother relationship quality; (3) father involvement (material support, in-kind support, direct father-child interaction); and (4) child outcomes (behavioral, social, emotional). The study will use an experimental design and randomly assign 180 AA fathers who are not currently involved with the criminal justice system and their 2-5 year old children to the BBTF or an attention control condition and assess outcomes at baseline, 12 weeks, and 24 weeks. Custodial mothers of the children will be recruited to concurrently complete child outcome measures, measures of father-mother relationship quality, and father involvement measures.

The specific aims and hypotheses are as follows:

Aim 1: Test the direct effects of the 9-session BBTF program on: (1) father's outcomes (psychological well-being, parenting competence, and communication and problem solving) and (2) paternal involvement (material support, in-kind support, and direct father-child interaction), controlling for father characteristics (demographics, history of criminal justice system involvement, social support) and child characteristics (age, gender). Hypothesis 1: BBTF program fathers will report better father outcomes and greater paternal involvement than the attention control group at 12 weeks and 24 weeks.

Aim 2: Test the mediating effects of father-mother relationship and father outcomes on paternal involvement across the two conditions. Hypothesis 2: Father-mother relationship quality and father outcomes will mediate intervention effects on paternal involvement.

Aim 3: Compare the effects of the BBTF program, controlling for father outcomes, father-mother relationship, and paternal involvement on child outcomes (behavioral, emotional/social development) as compared to the attention control group. Hypothesis 3a: BBTF children will have improved child outcomes relative to the control group at 12 weeks and 24 weeks. Hypothesis 3b: Child outcomes will be mediated by improvements in father outcomes, paternal involvement and father-mother relationship.

ELIGIBILITY:
Inclusion Criteria:

* AA biological father of a child 2 to 5 years old
* Child lives with father no more than 48 hours per week (e.g., spends the weekends with his or her father)
* The child lives with the biological mother (or other custodial relative such as grandmother) in the metropolitan Chicago area.
* These fathers are referred to as AA non-resident fathers. Additional criteria include: (1) child's mother is willing to consent to complete the child assessments; - Child's mother is amenable to facilitating opportunities for fathers to interact with their children in order to practice skills learned in the program
* Father is able and willing to travel to one of two intervention sites to attend a weekly program.
* The study is limited to fathers with a target child aged 2-5 years.
* The rationale for this limit is based on the developmental phase when families are most vulnerable to decreased father involvement and children are highly dependent on parenting for their growth and development.

Exclusion Criteria:

* Fathers with histories of child abuse, neglect, or violence perpetuated against the child or the child's mother (based on mother or father report).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 308 (Actual)
Dates: Start 2015-02; Primary Completion 2018-09-24 (Actual); Study Completion 2018-09-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wrenetha Julion, PhD, Principal Investigator — Rush University
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

REFERENCES:
- [Background] Julion WA, Breitenstein SM, Waddell D. Fatherhood intervention development in collaboration with African American non-resident fathers. Res Nurs Health. 2012 Oct;35(5):490-506. doi: 10.1002/nur.21492. Epub 2012 Jun 8. PMID 22685066
- [Background] Julion W, Gross D, Barclay-McLaughlin G, Fogg L. "It's not just about MOMMAS": African-American non-resident fathers' views of paternal involvement. Res Nurs Health. 2007 Dec;30(6):595-610. doi: 10.1002/nur.20223. PMID 18022813
- [Result] Julion WA, Sumo J, Bounds DT, Breitenstein SM, Schoeny M, Gross D, Fogg L. Study protocol for a randomized clinical trial of a fatherhood intervention for African American non-resident fathers: Can we improve father and child outcomes? Contemp Clin Trials. 2016 Jul;49:29-39. doi: 10.1016/j.cct.2016.05.005. Epub 2016 May 28. PMID 27241687
- [Result] Julion WA, Sumo J, Bounds DT. A tripartite model for recruiting African-Americans into fatherhood intervention research. Public Health Nurs. 2018 Sep;35(5):420-426. doi: 10.1111/phn.12411. Epub 2018 May 9. PMID 29740854
- [Result] Julion W, Sumo J, Schoeny ME, Breitenstein SM, Bounds DT. Recruitment, Retention, and Intervention Outcomes from the Dedicated African American Dad (DAAD) Study. J Urban Health. 2021 Oct;98(Suppl 2):133-148. doi: 10.1007/s11524-021-00549-8. Epub 2021 Jul 1. PMID 34196905

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Active and passive recruitment strategies were used.. Active approaches included meeting directly with potential participants or individuals who may know potential participants. Passive recruitment included providing study information without direct contact with members of the study team (i.e. by study advertisement and/or word of mouth recruitment efforts such as notices placed in church bulletins, neighborhood newsletters, community organizations' email blasts and live radio interviews).
Pre-assignment Details: Approximately 2 weeks prior to the start of the groups, participants were block randomized into the two conditions using the wave/cohort as a block. Microsoft Excel was used to randomly assign participants to the two groups. Fathers were randomized when consenting and baseline data collection had occurred. The requirement for imminent maternal data collection was removed in order to allow father participation in the study even if the mother was unwilling to provide data.
Period: Overall Study
Arm/Group | Financial Literacy Program | BBTF Intervention
Started | 145 | 163
Completed | 107 | 124
Not Completed | 38 | 39
Not completed — Lost to Follow-up | 38 | 39

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Financial Literacy Program | BBTF Intervention | Total
Number analyzed (Participants) | 145 | 163 | 308
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Missing cases did not report a valid date of birth. Fathers and Mothers are presented separately.
  years
    Age - Fathers: number analyzed (Participants) | 86 | 92 | 178
    Age - Fathers | 34.2 (8.9) | 33.0 (9.1) | 33.5 (9.0)
    Age - Mothers: number analyzed (Participants) | 58 | 69 | 127
    Age - Mothers | 31.6 (7.2) | 31.2 (7.1) | 31.4 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 71 | 130
  Male | 86 | 92 | 178
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Fathers and Mothers are presented separately.
  Participants
    Ethnicity - Fathers: number analyzed (Participants) | 86 | 92 | 178
    Ethnicity - Fathers: Hispanic or Latino | 6 | 4 | 10
    Ethnicity - Fathers: Not Hispanic or Latino | 80 | 87 | 167
    Ethnicity - Fathers: Unknown or Not Reported | 0 | 1 | 1
    Ethnicity - Mothers: number analyzed (Participants) | 59 | 71 | 130
    Ethnicity - Mothers: Hispanic or Latino | 0 | 1 | 1
    Ethnicity - Mothers: Not Hispanic or Latino | 37 | 43 | 80
    Ethnicity - Mothers: Unknown or Not Reported | 22 | 27 | 49
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Fathers and Mothers are presented separately.
  Participants
    Race - Fathers: number analyzed (Participants) | 86 | 92 | 178
    Race - Fathers: American Indian or Alaska Native | 0 | 0 | 0
    Race - Fathers: Asian | 0 | 0 | 0
    Race - Fathers: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Race - Fathers: Black or African American | 86 | 92 | 178
    Race - Fathers: White | 0 | 0 | 0
    Race - Fathers: More than one race | 0 | 0 | 0
    Race - Fathers: Unknown or Not Reported | 0 | 0 | 0
    Race - Mothers: number analyzed (Participants) | 59 | 71 | 130
    Race - Mothers: American Indian or Alaska Native | 3 | 0 | 3
    Race - Mothers: Asian | 0 | 0 | 0
    Race - Mothers: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Race - Mothers: Black or African American | 34 | 43 | 77
    Race - Mothers: White | 0 | 0 | 0
    Race - Mothers: More than one race | 0 | 0 | 0
    Race - Mothers: Unknown or Not Reported | 22 | 28 | 50
Marital Status [Count of Participants; unit: Participants] — Population: Fathers and Mothers are presented separately.
  Participants
    Marital Status - Fathers: number analyzed (Participants) | 86 | 92 | 178
    Marital Status - Fathers: Married or Living with a Domestic Partner | 1 | 5 | 6
    Marital Status - Fathers: Separated | 12 | 10 | 22
    Marital Status - Fathers: Divorced | 12 | 9 | 21
    Marital Status - Fathers: Never Married | 61 | 68 | 129
    Marital Status - Fathers: Missing/Not Reported | 0 | 0 | 0
    Marital Status - Mothers: number analyzed (Participants) | 59 | 71 | 130
    Marital Status - Mothers: Married or Living with a Domestic Partner | 5 | 3 | 8
    Marital Status - Mothers: Separated | 7 | 2 | 9
    Marital Status - Mothers: Divorced | 4 | 7 | 11
    Marital Status - Mothers: Never Married | 42 | 58 | 100
    Marital Status - Mothers: Missing/Not Reported | 1 | 1 | 2
Education Level [Count of Participants; unit: Participants] — Population: Fathers and Mothers are presented separately.
  Participants
    Education Level - Fathers: number analyzed (Participants) | 86 | 92 | 178
    Education Level - Fathers: High School Graduate or Less | 38 | 43 | 81
    Education Level - Fathers: Some College or More | 48 | 49 | 97
    Education Level - Fathers: Unknown/Not Reported | 0 | 0 | 0
    Education Level - Mothers: number analyzed (Participants) | 59 | 71 | 130
    Education Level - Mothers: High School Graduate or Less | 18 | 22 | 40
    Education Level - Mothers: Some College or More | 40 | 48 | 88
    Education Level - Mothers: Unknown/Not Reported | 1 | 1 | 2
Job/Employment Status [Count of Participants; unit: Participants] — Population: Fathers and Mothers are presented separately.
  Participants
    Job/Employment Status - Fathers: number analyzed (Participants) | 86 | 92 | 178
    Job/Employment Status - Fathers: Part Time | 22 | 21 | 43
    Job/Employment Status - Fathers: Full Time | 28 | 30 | 58
    Job/Employment Status - Fathers: Not Currently Working | 31 | 33 | 64
    Job/Employment Status - Fathers: Going to School | 2 | 3 | 5
    Job/Employment Status - Fathers: Working and Going to School | 3 | 5 | 8
    Job/Employment Status - Fathers: Unknown/Not Reported | 0 | 0 | 0
    Job/Employment Status - Mothers: number analyzed (Participants) | 59 | 71 | 130
    Job/Employment Status - Mothers: Part Time | 6 | 9 | 15
    Job/Employment Status - Mothers: Full Time | 31 | 34 | 65
    Job/Employment Status - Mothers: Not Currently Working | 11 | 16 | 27
    Job/Employment Status - Mothers: Going to School | 4 | 3 | 7
    Job/Employment Status - Mothers: Working and Going to School | 6 | 8 | 14
    Job/Employment Status - Mothers: Unknown/Not Reported | 1 | 1 | 2
Monthly Income [Count of Participants; unit: Participants] — Population: Fathers and Mothers are presented separately.
  Participants
    Monthly Income - Fathers: number analyzed (Participants) | 86 | 92 | 178
    Monthly Income - Fathers: $500 or less | 20 | 27 | 47
    Monthly Income - Fathers: $501-1000 | 19 | 18 | 37
    Monthly Income - Fathers: $1001-2000 | 22 | 24 | 46
    Monthly Income - Fathers: $2001-3000 | 6 | 10 | 16
    Monthly Income - Fathers: $3000 or more | 18 | 13 | 31
    Monthly Income - Fathers: Unknown/Not Reported | 1 | 0 | 1
    Monthly Income - Mothers: number analyzed (Participants) | 59 | 71 | 130
    Monthly Income - Mothers: $500 or less | 6 | 7 | 13
    Monthly Income - Mothers: $501-1000 | 11 | 21 | 32
    Monthly Income - Mothers: $1001-2000 | 23 | 18 | 41
    Monthly Income - Mothers: $2001-3000 | 12 | 12 | 24
    Monthly Income - Mothers: $3000 or more | 5 | 7 | 12
    Monthly Income - Mothers: Unknown/Not Reported | 2 | 6 | 8

OUTCOME MEASURES:

1. Primary Outcome: Father Involvement as Measured by the Fragile Families Survey - Father Report
Description: The Fragile Families Survey (FFS) Measures the frequency with which fathers provide material and in-kind support and directly interact with their child The minimum score is 13, and the maximum score is 52. Higher scores mean a better outcome.
Time Frame: Mean/Standard Error (SE) at Baseline, 12, and 24 weeks
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Financial Literacy Program - Fathers: The Financial Literacy Program (FLP) attention control condition will not receive any information on fatherhood. They will participate in a nine-session financial education program, called "Money Smart," which has modules that will be facilitated by a group leader that focus on banking, borrowing, checking accounts, money management, saving, establishing and repairing a credit history, using credit cards responsibly and learning about borrowing and home ownership. They will also receive a booster session 6 weeks after the final session that focuses on setting financial goals.
  Financial Literacy Program: The Financial Literacy Program (FLP) attention control condition consists of 9 group sessions and 1 booster session as described in the arm/group descriptions.
- BBTF Intervention - Fathers: The Building Bridges to Fatherhood (BBTF) intervention employs the following key features: a collaborative model for working with parents; vignettes of father-child models engaged in situations typical of non-resident fathers with young children for stimulating discussion and problem-solving; group discussion format, which allows fathers to support one another and share ideas on using program principles to fit within the contexts of fatherhood; "homework assignments" that help fathers practice the new skills at home; weekly handouts summarizing the major points discussed each week, which can be shared with others and used to gain greater support from extended family; and a Leader's Manual that standardizes the program across groups and group leaders.
  BBTF Intervention: The Building Bridges to Fatherhood (BBTF) intervention consists of 9 group sessions and 1 booster session as described in the arm/group descriptions.
Arm/Group | Financial Literacy Program - Fathers | BBTF Intervention - Fathers
Number analyzed (Participants) | 86 | 92
score on a scale
  Baseline | 41.1 (0.7) | 41.2 (0.7)
  12 Weeks | 41.6 (1.4) | 41.3 (1.6)
  24 Weeks | 41.5 (1.1) | 41.7 (1.1)
Statistical Analysis 1: Comparison: Financial Literacy Program - Fathers vs BBTF Intervention - Fathers; Data were analyzed using a 3 × 2 repeated measures analysis of covariance (RM-ANCOVA) with 3 assessments crossed with two treatment conditions (BBTF and FLP). Five variables were included as covariates: father's age, father's highest level of education, number of members in father's social network, number of adults in the household, and sex of the target child. The effect of interest was the condition x time interaction; Test type: Superiority; p = .962, ANCOVA

2. Primary Outcome: Father Involvement as Measured by the Julion Index of Paternal Involvement - Father Report
Description: The Julion Index of Paternal Involvement (JIPI) measured the frequency with which fathers provide material and in-kind support and engage in direct father-child interaction.
  The minimum value is 19 and the maximum value is 76. Higher scores mean a better outcome.
Time Frame: Change from baseline to 12 and 24 weeks
Population: This is a father-reported measure. Only fathers are reported in this analysis.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Financial Literacy Program - Fathers | BBTF Intervention - Fathers
Number analyzed (Participants) | 86 | 92
score on a scale
  Baseline | 66.4 (1.0) | 66.4 (1.1)
  12 Weeks | 65.0 (2.0) | 65.3 (2.0)
  24 Weeks | 68.5 (1.3) | 68.3 (1.2)
Statistical Analysis 1: Comparison: Financial Literacy Program - Fathers vs BBTF Intervention - Fathers; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .982, ANCOVA

3. Secondary Outcome: Taylor Inventory of Self-Esteem (Positive)
Description: The 16-item Taylor Inventory of Self-esteem is a measure of self-esteem and rewards and costs to self. The minimum value on the 8-item positive subscale is zero, and the maximum value is 64. Higher scores are better outcomes.
Time Frame: Mean/SE at Baseline, 12, and 24 weeks
Population: This is a father-reported measure. Only fathers are reported in this analysis.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Financial Literacy Program - Fathers | BBTF Intervention - Fathers
Number analyzed (Participants) | 86 | 92
score on a scale
  Baseline | 52.7 (0.8) | 54.3 (0.7)
  12 Weeks | 54.2 (1.5) | 53.6 (1.6)
  24 Weeks | 54.4 (1.0) | 54.3 (1.1)
Statistical Analysis 1: Comparison: Financial Literacy Program - Fathers vs BBTF Intervention - Fathers; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .534, ANCOVA

4. Secondary Outcome: Taylor Inventory of Self-Esteem (Negative)
Description: The 16-item Taylor Inventory of Self-esteem is a measure of self-esteem and rewards and costs to self. The minimum value on the 8-item negative subscale is zero, and the maximum value is 64. Higher scores are worse outcomes.
Time Frame: Baseline, 12, and 24 weeks
Population: This is a father-reported measure. Only fathers are reported in this analysis.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Financial Literacy Program - Fathers | BBTF Intervention - Fathers
Number analyzed (Participants) | 86 | 92
score on a scale
  Baseline | 38.1 (1.5) | 37.0 (1.6)
  12 Weeks | 40.2 (2.6) | 40.6 (2.3)
  24 Weeks | 41.2 (2.1) | 39.1 (1.8)
Statistical Analysis 1: Comparison: Financial Literacy Program - Fathers vs BBTF Intervention - Fathers; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .730, ANCOVA

5. Secondary Outcome: Perceived Stress Scale (Negative)
Description: The Perceived Stress Scale examines the degree to which situations are experienced as stressful. The 6-item negative subscale has a range of scores from zero to 24. Higher scores are worse outcomes.
Time Frame: Baseline, 12, and 24 weeks
Population: This is a father-reported measure. Only fathers are reported in this analysis.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Financial Literacy Program - Fathers | BBTF Intervention - Fathers
Number analyzed (Participants) | 86 | 92
score on a scale
  Baseline | 11.0 (.6) | 11.6 (.5)
  12 Weeks | 9.5 (1.1) | 9.9 (1.0)
  24 Weeks | 9.4 (.7) | 10.4 (.7)
Statistical Analysis 1: Comparison: Financial Literacy Program - Fathers vs BBTF Intervention - Fathers; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .927, ANCOVA

6. Secondary Outcome: Perceived Stress Scale (Positive)
Description: The Perceived Stress Scale examines the degree to which situations are experienced as stressful. The 4-item positive subscale has a range of scores from zero to 16. Higher scores are better outcomes.
Time Frame: Baseline, 12, and 24 weeks
Population: This is a father-reported measure. Only fathers are reported in this analysis.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Financial Literacy Program - Fathers | BBTF Intervention - Fathers
Number analyzed (Participants) | 86 | 92
score on a scale
  Baseline | 5.3 (.2) | 5.5 (.3)
  12 Weeks | 4.8 (.6) | 5.0 (.5)
  24 Weeks | 4.0 (.4) | 4.6 (.4)
Statistical Analysis 1: Comparison: Financial Literacy Program - Fathers vs BBTF Intervention - Fathers; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .841, ANCOVA

7. Secondary Outcome: Center for Epidemiologic Studies Depression Scale
Description: The Center for Epidemiologic Studies Depression Scale (CESD) measures depressive symptoms experienced in the past week.
  The minimum value is zero and the maximum value is sixty. Four items were reverse coded and higher scores indicated worse outcomes.
Time Frame: Baseline, 12, and 24 weeks
Population: This is a father-reported measure. Only fathers are reported in this analysis.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Financial Literacy Program - Fathers | BBTF Intervention - Fathers
Number analyzed (Participants) | 86 | 92
score on a scale
  Baseline | 13.7 (.9) | 14.9 (.9)
  12 Weeks | 13.6 (1.8) | 15.2 (1.8)
  24 Weeks | 12.5 (1.5) | 15.6 (1.4)
Statistical Analysis 1: Comparison: Financial Literacy Program - Fathers vs BBTF Intervention - Fathers; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .722, ANCOVA

8. Secondary Outcome: Parenting Sense of Competence Scale (Satisfaction)
Description: The Parent Sense of Competency Scale measures satisfaction and self-efficacy in their parenting role. The 9-item satisfaction subscale has a range of scores from nine to fifty-four. Higher scores are better parenting self-esteem.
Time Frame: Baseline, 12, and 24 weeks
Population: This is a father-reported measure. Only fathers are reported in this analysis.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Financial Literacy Program - Fathers | BBTF Intervention - Fathers
Number analyzed (Participants) | 86 | 92
score on a scale
  Baseline | 23.2 (.8) | 24.9 (.8)
  12 Weeks | 22.1 (1.4) | 23.2 (1.3)
  24 Weeks | 22.8 (1.4) | 22.9 (1.1)
Statistical Analysis 1: Comparison: Financial Literacy Program - Fathers vs BBTF Intervention - Fathers; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .715, ANCOVA

9. Secondary Outcome: Parenting Sense of Competence Scale (Self-Efficacy)
Description: The Parent Sense of Competency Scale measures satisfaction and self-efficacy in their parenting role. The 7-item self-efficacy subscale has a range of scores from seven to 42. Higher scores are better parenting self-esteem.
Time Frame: Baseline, 12, and 24 weeks
Population: This is a father-reported measure. Only fathers are reported in this analysis.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Financial Literacy Program - Fathers | BBTF Intervention - Fathers
Number analyzed (Participants) | 86 | 92
score on a scale
  Baseline | 14.5 (.6) | 14.4 (.6)
  12 Weeks | 15.1 (1.0) | 15.5 (1.0)
  24 Weeks | 14.7 (1.0) | 15.3 (.9)
Statistical Analysis 1: Comparison: Financial Literacy Program - Fathers; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .900, ANCOVA

10. Secondary Outcome: Parent Behavior Checklist (Discipline)
Description: The Parent Behavior Checklist is a measure of parenting skills and knowledge. The 10-item discipline subscale has a range of values from 1 to 4. This scale was log transformed, making the range 0 to 1.4. Higher scores mean worse outcomes.
Time Frame: Baseline, 12, and 24 weeks
Population: This is a father-reported measure. Only fathers are reported in this analysis.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Financial Literacy Program - Fathers | BBTF Intervention - Fathers
Number analyzed (Participants) | 86 | 92
score on a scale
  Baseline | .37 (.03) | .35 (.02)
  12 Weeks | .38 (.05) | .31 (.04)
  24 Weeks | .33 (.04) | .37 (.04)
Statistical Analysis 1: Comparison: Financial Literacy Program - Fathers vs BBTF Intervention - Fathers; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .271, ANCOVA

11. Secondary Outcome: Parent Behavior Checklist (Nurturing)
Description: The Parent Behavior Checklist is a measure of parenting skills and knowledge. The 10-item nurturing subscale has a range of values from 1 to 4. Higher scores mean worse outcomes.
Time Frame: Baseline, 12, and 24 weeks
Population: This is a father-reported measure. Only fathers are reported in this analysis.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Financial Literacy Program - Fathers | BBTF Intervention - Fathers
Number analyzed (Participants) | 86 | 92
score on a scale
  Baseline | 3.0 (.05) | 3.0 (.05)
  12 Weeks | 3.1 (.1) | 3.1 (.1)
  24 Weeks | 3.1 (.1) | 3.1 (.1)
Statistical Analysis 1: Comparison: Financial Literacy Program - Fathers vs BBTF Intervention - Fathers; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .987, ANCOVA

12. Secondary Outcome: Parent Behavior Checklist (Expectations)
Description: The Parent Behavior Checklist is a measure of parenting skills and knowledge. The 12-item expectations subscale has a range of values from 1 to 4. Higher scores mean worse outcomes.
Time Frame: Baseline, 12, and 24 weeks
Population: This is a father-reported measure. Only fathers are reported in this analysis.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Financial Literacy Program - Fathers | BBTF Intervention - Fathers
Number analyzed (Participants) | 86 | 92
score on a scale
  Baseline | 3.1 (.1) | 3.0 (.1)
  12 Weeks | 3.1 (.1) | 3.1 (.1)
  24 Weeks | 3.3 (.1) | 3.2 (.1)
Statistical Analysis 1: Comparison: Financial Literacy Program - Fathers vs BBTF Intervention - Fathers; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .967, ANCOVA

13. Secondary Outcome: Quality of Relationship Inventory (Support)
Description: Measure of support, conflict, and depth of father-mother relationship. The Quality of Relationship Inventory (QRI) a self-assessment questionnaire used to determine the quality of a couple's relationship and their satisfaction with the relationship. The minimum score on the support subscale is 1 and the maximum score is 4. Higher scores mean a better outcome.
Time Frame: Baseline, 12, and 24 weeks
Population: This is a father-reported measure. Only fathers are reported in this analysis.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Financial Literacy Program - Fathers | BBTF Intervention - Fathers
Number analyzed (Participants) | 86 | 92
score on a scale
  Baseline | 2.5 (.1) | 2.4 (.1)
  12 Weeks | 2.5 (.2) | 2.5 (.2)
  24 Weeks | 2.4 (.1) | 2.5 (.1)
Statistical Analysis 1: Comparison: Financial Literacy Program - Fathers vs BBTF Intervention - Fathers; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .693, ANCOVA

14. Secondary Outcome: Quality of Relationship Inventory (Conflict)
Description: Measure of support, conflict, and depth of father-mother relationship. The Quality of Relationship Inventory (QRI) a self-assessment questionnaire used to determine the quality of a couple's relationship and their satisfaction with the relationship. The minimum score on the conflict subscale is 1and the maximum score is 4. Higher scores mean a worse outcome..
Time Frame: Baseline, 12, and 24 weeks
Population: This is a father-reported measure. Only fathers are reported in this analysis.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Financial Literacy Program - Fathers | BBTF Intervention - Fathers
Number analyzed (Participants) | 86 | 92
score on a scale
  Baseline | 2.5 (.1) | 2.5 (.1)
  12 Weeks | 2.2 (.1) | 2.3 (.1)
  24 Weeks | 2.4 (.1) | 2.3 (.1)
Statistical Analysis 1: Comparison: Financial Literacy Program - Fathers vs BBTF Intervention - Fathers; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .557, ANCOVA

15. Secondary Outcome: Quality of Relationship Inventory (Depth)
Description: Measure of support, conflict, and depth of father-mother relationship. The Quality of Relationship Inventory (QRI) a self-assessment questionnaire used to determine the quality of a couple's relationship and their satisfaction with the relationship. The minimum score on the depth subscale is 1 and the maximum score is 4. Higher scores mean a better outcome.
Time Frame: Baseline, 12, and 24 weeks
Population: This is a father-reported measure. Only fathers are reported in this analysis.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Financial Literacy Program - Fathers | BBTF Intervention - Fathers
Number analyzed (Participants) | 86 | 92
score on a scale
  Baseline | 2.6 (.1) | 2.4 (.1)
  12 Weeks | 2.5 (.2) | 2.4 (.2)
  24 Weeks | 2.5 (.1) | 2.4 (.1)
Statistical Analysis 1: Comparison: Financial Literacy Program - Fathers vs BBTF Intervention - Fathers; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .681, ANCOVA

16. Secondary Outcome: Behavior Assessment System for Children 3rd Ed (Aggression)
Description: The Behavior Assessment System for Children (BASC) is a measure of adaptive and problem behaviors in community and home settings. The aggression subscale measures the tendency to act in a hostile manner (either verbal or physical) that is threatening to others. The raw scores are converted to T-Scores with a population mean of 50 and standard deviation of 10. Higher scores mean a worse outcome. Scores 70 and above are considered clinically significant level.
Time Frame: Baseline, 12, and 24 weeks
Population: This is a father-reported measure. Only fathers are reported in this analysis.
Measure: Mean (Standard Error); unit: T scores
Arm/Group | Financial Literacy Program - Fathers | BBTF Intervention - Fathers
Number analyzed (Participants) | 86 | 92
T scores
  Baseline | 49.0 (1.2) | 46.8 (1.0)
  12 Weeks | 47.3 (2.3) | 48.7 (2.3)
  24 Weeks | 51.1 (2.2) | 53.0 (2.2)
Statistical Analysis 1: Comparison: Financial Literacy Program - Fathers vs BBTF Intervention - Fathers; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .389, ANCOVA

17. Secondary Outcome: Behavior Assessment System for Children 3rd Ed (Attention)
Description: The Behavior Assessment System for Children (BASC) is a measure of adaptive and problem behaviors in community and home settings. The attention subscale measures he tendency to be easily distracted and unable to concentrate more than momentarily. The raw scores are converted to T-Scores with a population mean of 50 and standard deviation of 10. Higher scores mean a worse outcome. Scores 70 and above are considered clinically significant level.
Time Frame: Baseline, 12, and 24 weeks
Population: This is a father-reported measure. Only fathers are reported in this analysis.
Measure: Mean (Standard Error); unit: T scores
Arm/Group | Financial Literacy Program - Fathers | BBTF Intervention - Fathers
Number analyzed (Participants) | 86 | 92
T scores
  Baseline | 49.4 (.9) | 51.0 (1.0)
  12 Weeks | 48.5 (2.0) | 48.5 (2.0)
  24 Weeks | 48.3 (1.7) | 48.6 (1.6)
Statistical Analysis 1: Comparison: Financial Literacy Program - Fathers vs BBTF Intervention - Fathers; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .846, ANCOVA

18. Secondary Outcome: Behavior Assessment System for Children 3rd Ed (Depression)
Description: The Behavior Assessment System for Children (BASC) is a measure of adaptive and problem behaviors in community and home settings. The depression subscale measures feelings of unhappiness, sadness, and stress that may result in an inability to carry out everyday activities or may bring on thoughts of suicide. The raw scores are converted to T-Scores with a population mean of 50 and standard deviation of 10. Higher scores mean a worse outcome. Scores 70 and above are considered clinically significant level.
Time Frame: Baseline, 12, and 24 weeks
Population: This is a father-reported measure. Only fathers are reported in this analysis.
Measure: Mean (Standard Error); unit: T scores
Arm/Group | Financial Literacy Program - Fathers | BBTF Intervention - Fathers
Number analyzed (Participants) | 86 | 92
T scores
  Baseline | 49.8 (1.2) | 50.2 (1.1)
  12 Weeks | 50.0 (2.8) | 51.5 (2.5)
  24 Weeks | 52.7 (2.1) | 52.3 (2.3)
Statistical Analysis 1: Comparison: Financial Literacy Program - Fathers vs BBTF Intervention - Fathers; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .871, ANCOVA

19. Secondary Outcome: Behavior Assessment System for Children 3rd Ed (Hyperactivity)
Description: The Behavior Assessment System for Children (BASC) is a measure of adaptive and problem behaviors in community and home settings. The hyperactivity subscale measures the tendency to be overly active, rush through work or activities, and act without thinking. The raw scores are converted to T-Scores with a population mean of 50 and standard deviation of 10. Higher scores mean a worse outcome. Scores 70 and above are considered clinically significant level.
Time Frame: Baseline, 12, and 24 weeks
Population: This is a father-reported measure. Only fathers are reported in this analysis.
Measure: Mean (Standard Error); unit: T scores
Arm/Group | Financial Literacy Program - Fathers | BBTF Intervention - Fathers
Number analyzed (Participants) | 86 | 92
T scores
  Baseline | 49.6 (1.1) | 49.9 (1.1)
  12 Weeks | 50.5 (2.4) | 50.8 (2.0)
  24 Weeks | 42.0 (1.9) | 51.8 (1.7)
Statistical Analysis 1: Comparison: Financial Literacy Program - Fathers vs BBTF Intervention - Fathers; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .986, ANCOVA

20. Secondary Outcome: Tolerance For Disagreement
Description: The degree of tolerance of interpersonal disagreement. The minimum score is 15 and the maximum score is 75. Higher scores mean a better outcome.
Time Frame: Baseline, 12, and 24 weeks
Population: This is a father-reported measure. Only fathers are reported in this analysis.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Financial Literacy Program - Fathers | BBTF Intervention - Fathers
Number analyzed (Participants) | 86 | 92
score on a scale
  Baseline | 41.0 (0.8) | 41.9 (0.8)
  12 Weeks | 39.5 (1.6) | 39.2 (1.5)
  24 Weeks | 41.1 (1.2) | 40.7 (1.3)
Statistical Analysis 1: Comparison: Financial Literacy Program - Fathers vs BBTF Intervention - Fathers; Test type: Superiority; p = .791, ANCOVA

21. Secondary Outcome: Personal Problem Solving Inventory - Efficacy
Description: The Perceived Problem Solving Inventory subscale measures perceived efficacy in one's own ability to solve problems. The minimum score is 1 and the maximum score is 6 for each of the 7 items. The total range of scores for this subscale is from 1 to 6. Higher scores mean a worse outcome.
Time Frame: Baseline, 12, and 24 weeks
Population: This is a father-reported measure. Only fathers are reported in this analysis.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Financial Literacy Program - Fathers | BBTF Intervention - Fathers
Number analyzed (Participants) | 86 | 92
score on a scale
  Baseline | 2.1 (0.1) | 2.1 (0.1)
  12 Weeks | 1.9 (0.1) | 1.7 (0.1)
  24 Weeks | 1.8 (0.1) | 1.9 (0.1)
Statistical Analysis 1: Comparison: Financial Literacy Program - Fathers vs BBTF Intervention - Fathers; Test type: Superiority; p = .583, ANCOVA

22. Secondary Outcome: Personal Problem Solving Inventory - Skills
Description: The Personal Problem Solving Inventory measures perceived skills in one's own ability to solve problems. The minimum score is 1 and the maximum score is 6 for each of the 9 items on this subscale. Total range of scores for the scale are 1 to 6. Higher scores mean a worse outcome.
Time Frame: Baseline, 12, and 24 weeks
Population: This is a father-reported measure. Only fathers are reported in this analysis.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Financial Literacy Program - Fathers | BBTF Intervention - Fathers
Number analyzed (Participants) | 86 | 92
score on a scale
  Baseline | 2.1 (0.1) | 2.1 (0.1)
  12 Weeks | 1.9 (0.1) | 1.8 (0.1)
  24 Weeks | 2.1 (0.1) | 2.0 (0.1)
Statistical Analysis 1: Comparison: Financial Literacy Program - Fathers vs BBTF Intervention - Fathers; Test type: Superiority; p = .851, ANCOVA

23. Other Pre Specified Outcome: Building Bridges To Fatherhood (BBTF) Social Context Validity
Description: An investigator developed Weekly Satisfaction and Program Satisfaction Survey was used to measure the levels of consumer satisfaction and active participation in the intervention. The 5-item weekly satisfaction survey minimum score is 0 and highest score is 15. The 16-item Program Satisfaction survey minimum score is 0 and the highest score is 48. Higher scores reflect greater satisfaction.
Time Frame: 9 weeks post baseline
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 36 months
Description: Adverse events were monitored over the 36 month time period but no adverse events were experienced by participants. There are only 2 arms in the study.
  Only fathers are reported in the analyses.
Arm/Group | Financial Literacy Program | BBTF Intervention
All-Cause Mortality (participants affected / at risk) | 0/86 | 0/92
Serious Adverse Events (participants affected / at risk) | 0/86 | 0/92
Other Adverse Events (participants affected / at risk) | 0/86 | 0/92

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (4):
  • Study Protocol and Statistical Analysis Plan (2016-07-15): https://cdn.clinicaltrials.gov/large-docs/48/NCT02412748/Prot_SAP_000.pdf
  • Informed Consent Form: ICF_Father (2018-07-07): https://cdn.clinicaltrials.gov/large-docs/48/NCT02412748/ICF_001.pdf
  • Informed Consent Form: ICF_Mother (2018-07-06): https://cdn.clinicaltrials.gov/large-docs/48/NCT02412748/ICF_002.pdf
  • Informed Consent Form: ICF_Mother_telephone consent (2018-07-06): https://cdn.clinicaltrials.gov/large-docs/48/NCT02412748/ICF_003.pdf